CLINICAL TRIAL: NCT05990205
Title: Effect of the Genetic Variants Typical of the Mestizo Population That Confer Risk of Having Metabolic Diseases on the Response to Common Treatments (Diet, Physical Activity, Metformin, Exercise).
Brief Title: Effect of the SCL16A11 Risk Haplotype on Treatments to Prevent Type 2 Diabetes
Acronym: PRED2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2579
Record Dates: First submitted 2023-07-18; First posted 2023-08-14 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2023-05

CONDITIONS: PreDiabetes
Keywords: PreDiabetes; Metformin; Precision nutrition; SLC16A11; Mexican Mestizos
MeSH Terms: conditions — Prediabetic State | interventions — Metformin; Laser Speckle Contrast Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Life Style Intervention (Active Comparator): Hypocaloric diet, 25 kcal/kg of ideal weight, 45% of the total intake of carbohydrates, 30% lipids, and 25% protein sources + physical activity (>150 min medium intensity per week)
  Interventions: Behavioral: Life Style Intervention
- Life Style Intervention + Metformin (Active Comparator): Hypocaloric diet, 25 kcal/kg of ideal weight, 45% of the total intake of carbohydrates, 30% lipids, and 25% protein sources + physical activity (>150 min medium intensity per week) + (750 mg metformin twice a day).
  Interventions: Drug: Life Style Intervention + Metformin

INTERVENTIONS:
Drug: Life Style Intervention + Metformin — hypocaloric diet, 25 kcal/kg of ideal weight, 45% of the total intake of carbohydrates, 30% lipids, and 25% protein sources + physical activity (>150 min medium intensity per week) + Metformin extended release 750mg each 12 hours
  Other Names: LSI + MET
  Arms: Life Style Intervention + Metformin
Behavioral: Life Style Intervention — hypocaloric diet, 25 kcal/kg of ideal weight, 45% of the total intake of carbohydrates, 30% lipids, and 25% protein sources + physical activity (>150 min medium intensity per week)
  Other Names: LSI
  Arms: Life Style Intervention

SUMMARY:
The goal of this randomized clinical trial is to determine the impact of the risk haplotype on SLC16A11 on early therapeutic responses in treatments to prevent T2D in Mexican mestizos with prediabetes. The main question[s] it aims to answer are:

* Evaluate the effect of the risk haplotype on weigth loss >3%
* Evualuate the differences in lipid profiles and glycemic parameters (fasting glucose, HbA1c).

Participants will be randomized into two groups: lifestyle intervention (LSI): hypocaloric diet, 25 kcal/kg of ideal weight, 45% of the total intake of carbohydrates, 30% lipids, and 25% protein sources + physical activity (>150 min medium intensity per week), or LSI + MET (750 mg metformin twice a day).

Researchers will compare carriers and non carriers of the risk haplotype of SLC16A11 to see if there are diferent treatment responses.

DETAILED DESCRIPTION:
Objectives: Dietary modification and/or metformin remain the most cost-effective treatment to prevent type 2 diabetes (T2D). Yet, there is an important variation in receiving the benefit among individuals. A haplotype in SLC16A11 is associated with decreased insulin action and risk for T2D in Mexicans. We aim to determine the impact of the risk haplotype on SLC16A11 on early therapeutic responses in treatments to prevent T2D.

Methods: We recrute individuals with at least one prediabetes criteria according to the American Diabetes Association with a body mass index (BMI) between 25 and 45 kg/m2. Participants are randomized into two groups: lifestyle intervention (LSI): hypocaloric diet, 25 kcal/kg of ideal weight, 45% of the total intake of carbohydrates, 30% lipids, and 25% protein sources + physical activity (>150 min medium intensity per week), or LSI + MET (750 mg metformin twice a day). Standardized dietitians delivere the LSI. The treatment goal is to achieve >3% weight loss during the 12-week follow-up. Participants are genotyped for the risk allele rs13342232 and rs75493593. The effects of the risk haplotype are evaluated with linear and logistic regressions adjusted by age, sex, five genetic principal components, BMI, and prediabetes criteria at baseline. Primary outcome is a significant interaction between the treatment arm and genotype in weight loss goal >3% after the treatment. Secondary outcome are differences in lipid levels and third outcome is differences in glycemic parameters (fasting glucose, HbA1c).

ELIGIBILITY:
Inclusion Criteria:

* Mexican mestizos
* At least one prediabetes criteria according to the American Diabetes Association: fasting glucose between 100-124 mg/dL, Glycosylated hemoglobin (HbA1c) between 5.7-6.4, and 2-hour blood sugar between 140 mg/dl-199 mg/dl after an oral load of 75g of glucose) (1);
* Age ranged between 18-65 years
* Overweight or obesity (BMI between 25.0 - 40 kg/m2).

Exclusion Criteria:

* Chronic diseases
* Pregnancy
* Chronic use of medications that altered plasma glucose levels.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Change in weigth loss | 12 weeks
  Number of participants in each treatment arm reaching the the goal weight loss >3%

SECONDARY OUTCOMES:
Change in Total-Cholesterol parameters | 12 weeks
  Decreasing concentration of Total-Cholesterol (mg/dl)
Change in LDL-Cholesterol parameters | 12 weeks
  Decreasing LDL-Cholesterol levels (mg/dl)
Change in ApoB | 12 weeks
  Decreasing ApoB levels (mg/dl)
Change in NonHDL-Cholesterol | 12 weeks
  Decreasin NonHDL-Cholesterol levels (mg/dl)
Change in fasting glucose | 12 weeks
  Decreasing fasting glucose levels (mg/dl)
Change in HbA1c | 12 weeks
  Decreasin HbA1c levels (%)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Aguilar Salinas, PhD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared upon request to authorized researchers
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available to the broader scientific community within six months of publication or within 18 months of the conclusion of the funding period if the study remains unpublished.
Access Criteria: Per International standards, we will require from any investigator or entity requesting the data a data-sharing agreement that provides (1) a commitment to using the data only for research purposes and not to identify any individual participants, (2) a commitment to securing the data using appropriate computer technology, and (3) a commitment to destroying or returning the data after analyses are completed.